CLINICAL TRIAL: NCT02815267
Title: A Randomized, Double-Blind Study to Compare the Efficacy, Safety and Long-Term Safety of Topical Administration of FMX-101 for 1 Year in the Treatment of Moderate-to-Severe Acne Vulgaris, Study FX2014-04
Brief Title: A Study to Compare the Efficacy and Safety of Topical Administration of FMX-101 for Treatment of Moderate-to-Severe Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FX2014-04
Record Dates: First submitted 2016-05-24; First posted 2016-06-28 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMX-101, 4% minocycline foam (Experimental): Subjects will apply the assigned FMX-101, 4% minocycline foam topically once daily for 12 weeks as directed
  Interventions: Drug: FMX-101, 4% minocycline foam
- Vehicle foam (Placebo Comparator): Subjects will apply the assigned vehicle foam topically once daily for 12 weeks as directed
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: FMX-101, 4% minocycline foam — FMX-101, 4% minocycline foam applied topically once daily for 12 weeks
  Arms: FMX-101, 4% minocycline foam
Drug: Vehicle Foam — Vehicle foam applied topically once daily for 12 weeks
  Arms: Vehicle foam

SUMMARY:
This is a Phase 3 study to evaluate the efficacy, safety and long-term safety of the topical administration of FMX-101, 4% minocycline foam for the treatment of moderate-to-severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Has facial acne vulgaris with:

  * 20 to 50 inflammatory lesions (papules, pustules, and nodules);
  * 25 to 100 noninflammatory lesions (open and closed comedones);
  * no more than 2 nodules on the face; and
  * IGA score of moderate (3) to severe (4)
* Willing to use only the supplied non-medicated cleanser (Cetaphil Gentle Skin Cleanser) and to refrain from use of any other acne medication, medicated cleanser, excessive sun exposure, and tanning booths for the duration of the study

Exclusion Criteria:

* Acne conglobata, acne fulminans, secondary acne (chloracne, drug induced acne) or any dermatological condition of the face or facial hair (eg, beard, sideburns, mustache) that could interfere with the clinical evaluations
* Sunburn on the face
* Severe systemic disease, which might interfere with the conduct of the study or the interpretation of the results.
* Abnormal baseline laboratory values that are considered clinically significant
* Allergy to tetracycline-class antibiotics or to any ingredient in the study drug
* Pseudomembranous colitis or antibiotic-associated colitis

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - Birmingham, Alabama
  - Fremont, California
  - Fullerton, California
  - Shelton, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Miami, Florida
  - Miramar, Florida
  - Sanford, Florida
  - Savannah, Georgia
  - Oakbrook Terrace, Illinois
  - Evansville, Indiana
  - Metairie, Louisiana
  - Rockville, Maryland
  - Bay City, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - New York, New York
  - High Point, North Carolina
  - Columbus, Ohio
  - Gresham, Oregon
  - Johnston, Rhode Island
  - Murfreesboro, Tennessee
  - Dallas, Texas
  - Plano, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Bridgeport, West Virginia
- San Cristóbal, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 35 sites in the United States and one site in the Dominican Republic from 06 May 2016 to 13 October 2017.
Pre-assignment Details: The study consisted of a varied screening period. All participants underwent inclusion and exclusion criteria assessment and all eligible participants signed the informed consent before undergoing any study related procedures. All assessments at screening were done as per the schedule of assessment.
Groups:
- FMX-101, 4% Minocycline Foam: Randomized participants applied FMX101 4% topically to the face once daily for 12 weeks as directed.
- Vehicle Foam: Randomized participants applied matching vehicle foam topically to the face once daily for 12 weeks as directed.
Period: Double-Blind Phase
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Started | 307 | 159
Completed | 274 | 128
Not Completed | 33 | 31
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 17 | 9
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Protocol Violation | 3 | 2
Not completed — Site withdrawal | 1 | 6
Not completed — Received a disallowed medication | 1 | 1
Period: Open-Label Phase
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Started | 193 | 91
Completed | 122 | 50
Not Completed | 71 | 41
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 23 | 9
Not completed — Withdrawal by Subject | 24 | 13
Not completed — Protocol Violation | 0 | 1
Not completed — Administrative | 21 | 12
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Population: Double-blind participants (Intent-to-Treat population) were moved to open-label (safety population)
Groups:
- Double-blind-FMX-101, 4% Minocycline Foam: Randomized participants applied FMX101 4% topically to the face once daily for 12 weeks as directed.
- Double-blind-Vehicle Foam: Randomized participants applied matching vehicle foam topically to the face once daily for 12 weeks as directed.
- Total: Total of all reporting groups
Arm/Group | Double-blind-FMX-101, 4% Minocycline Foam | Double-blind-Vehicle Foam | Total
Number analyzed (Participants) | 307 | 159 | 466
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.5 (7.5) | 20.0 (8.1) | 20.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 98 | 266
  Male | 139 | 61 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 36 | 112
  Not Hispanic or Latino | 231 | 123 | 354
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 10 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 86 | 40 | 126
  White | 192 | 100 | 292
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in the Inflammatory Lesion Count at Week 12
Description: To evaluate the efficacy in the treatment of acne compared to vehicle of topical FMX101 4% administered daily for 12 weeks. Changes from Baseline are calculated as Baseline value minus post-Baseline value, so that decreases appear as positive values. Inflammatory lesion count included: papules, pustules, and nodules.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) population: included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 307 | 159
Lesion counts | 13.95 (0.65) | 11.15 (0.90)
Statistical Analysis 1: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Change from baseline in inflammatory lesion count was analyzed using an analysis of covariance (ANCOVA) model, which included treatment, Baseline inflammatory lesion count and pooled investigational site as a blocking factor; Test type: Superiority; p = 0.0083, ANCOVA; Mean Difference (Final Values) = 2.80, 95% CI 2-sided [0.72 to 4.88], Standard Error of Mean 1.06

2. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessments (IGA) Treatment Success at Week 12
Description: The IGA scale for acne vulgaris, was used by the investigators to assess the severity of a participant's acne vulgaris. The scale ranges from 0 (Clear): normal, clear skin with no evidence of acne vulgaris to 5 (Very Severe): highly inflammatory lesions predominate, variable number of comedones, many papules/pustules and many nodulocystic lesions. Higher scores indicated severe outcome. Treatment success was defined as an IGA score of 0 (score of clear) or 1 (almost clear), and at least a 2-grade improvement (decrease) from Baseline.
Time Frame: Baseline and Week 12
Population: An ITT population: included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 307 | 159
Percentage of participants | 8.09 | 4.77
Statistical Analysis 1: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority; p = 0.1805, Cochran-Mantel-Haenszel — P-value is for the null hypothesis that the combined risk difference equals 0; Risk Difference (RD) = 3.33, 95% CI 2-sided [-1.54 to 8.19], Standard Error of Mean 2.48

3. Secondary Outcome: Percent Change From Baseline in the Non-inflammatory Lesion Count at Week 12
Description: To evaluate the efficacy in the treatment of acne compared to vehicle of topical FMX101 4% administered daily for 12 weeks. Percent change from Baseline is calculated as the Baseline value minus the post-Baseline value divided by the baseline value, expressed as a percentage. Non-inflammatory lesions included: open comedones (blackhead) and closed comedones (whitehead).
Time Frame: Baseline and Week 12
Population: An ITT Population: included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 307 | 159
Lesion counts | 32.34 (2.64) | 19.60 (3.81)
Statistical Analysis 1: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority — Percent change from baseline was analyzed using an ANCOVA model, which included treatment, baseline non-inflammatory lesion counts and pooled investigational site as a blocking factor. For the superiority comparison between FMX101 4% and vehicle; p = 0.0040, ANCOVA; Mean Difference (Final Values) = 12.73, 95% CI 2-sided [4.07 to 21.39], Standard Error of Mean 4.42

4. Secondary Outcome: Absolute Change From Baseline in the Inflammatory Lesion Count at Week 6 and Week 9
Description: as for outcome 1
Time Frame: Baseline, at Week 6 and at Week 9
Population: An ITT population: included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Lesion counts
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 307 | 159
Lesion counts
  Week 6 | 11.65 (0.63) | 7.79 (0.87)
  Week 9 | 13.24 (0.63) | 8.85 (0.87)
Statistical Analysis 1: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority — Change from baseline in inflammatory lesion count for Week 6 was analyzed using an ANCOVA model, which included treatment, baseline inflammatory lesion counts and pooled investigational site as a blocking factor; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 3.86, 95% CI 2-sided [1.85 to 5.87], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority — Change from baseline in inflammatory lesion count for Week 9 was analyzed using an ANCOVA model, which included treatment, baseline inflammatory lesion counts and pooled investigational site as a blocking factor; p < .0001, ANCOVA; Mean Difference (Final Values) = 4.39, 95% CI 2-sided [2.38 to 6.40], Standard Error of Mean 1.03

5. Secondary Outcome: Percentage of Participants Achieving IGA Treatment Success at Week 6 and Week 9
Description: as for outcome 2
Time Frame: Baseline, at Week 6 and at Week 9
Population: An ITT population: included all randomized population.
Measure: Number; unit: Percentage of participants
Arm/Group | FMX-101, 4% Minocycline Foam | Vehicle Foam
Number analyzed (Participants) | 307 | 159
Percentage of participants
  Week 6 | 3.47 | 0.75
  Week 9 | 4.19 | 1.43
Statistical Analysis 1: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority — P-value is for null hypothesis that the combined risk difference equals 0. Percentage of participants achieving IGA treatment success at Week 6; p = 0.0395, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.71, 95% CI 2-sided [0.13 to 5.3], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: FMX-101, 4% Minocycline Foam vs Vehicle Foam; Test type: Superiority — P-value is for null hypothesis that the combined risk difference equals 0. Percentage of participants achieving IGA treatment success at Week 9; p = 0.0748, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.76, 95% CI 2-sided [-0.28 to 5.80], Standard Error of Mean 1.55

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and and Treatment-emergent Serious Adverse Events (TESAEs)
Description: To evaluate the safety compared to vehicle of topical FMX101 4% administered daily for 12 weeks and to evaluate the long-term safety of topical FMX101 4% administered daily for up to an additional 40 weeks. TEAEs of the double-blind phase were defined as AEs starting on or after date of first application of investigational product (IP), but before the date of the first application of the open-label phase, and AEs starting on or after the first application of the open-label phase are considered as TEAEs of the open-label phase.
Time Frame: Double blind: Screening Day until Week 12; Open-label: Week 16 until Week 52
Population: Safety population: included all randomized participants who received IP. Participants who had no post-Baseline assessments were included in the Safety population unless all dispensed IP was returned unused.
Measure: Count of Participants; unit: Participants
Groups:
- Open-label-FMX-101, 4% Minocycline Foam: Selected participants from double-blind period received FMX101 4% minocycline foam for additional 40 weeks as directed in open-label period.
Arm/Group | Double-blind-FMX-101, 4% Minocycline Foam | Double-blind-Vehicle Foam | Open-label-FMX-101, 4% Minocycline Foam
Number analyzed (Participants) | 307 | 159 | 284
Participants
  Any TEAE | 52 | 29 | 65
  Any Treatment-related TEAE | 6 | 4 | 5
  Any Serious TEAE | 1 | 0 | 1
  Any TEAE Leading to IP Discontinuation | 0 | 3 | 2

ADVERSE EVENTS:
Time Frame: Double blind: Screening Day until Week 12; Open-label: Week 16 until Week 52
Arm/Group | Double-blind-FMX-101, 4% Minocycline Foam | Double-blind-Vehicle Foam | Open-label-FMX-101, 4% Minocycline Foam
All-Cause Mortality (participants affected / at risk) | 0/307 | 0/159 | 0/284
Serious Adverse Events (participants affected / at risk) | 1/307 | 0/159 | 1/284
Other Adverse Events (participants affected / at risk) | 13/307 | 11/159 | 19/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind-FMX-101, 4% Minocycline Foam (N=307) | Double-blind-Vehicle Foam (N=159) | Open-label-FMX-101, 4% Minocycline Foam (N=284)
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind-FMX-101, 4% Minocycline Foam (N=307) | Double-blind-Vehicle Foam (N=159) | Open-label-FMX-101, 4% Minocycline Foam (N=284)
Nasopharyngitis (Infections and infestations) | 6 | 6 | 10
Headache (Nervous system disorders) | 7 | 5 | 4
Influenza (Infections and infestations) | 0 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02815267/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT02815267/SAP_001.pdf